CLINICAL TRIAL: NCT06753890
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Clinical Trial, Efficacy and Safety Study of Changkang Granules in the Treatment of Irritable Bowel Syndrome With Predominant Diarrhea ( Liver qi Affecting the Spleen Pattern)
Brief Title: Efficacy and Safety of Changkang Granules in the Treatment of Irritable Bowel Syndrome With Predominant Diarrhea (Liver qi Affecting the Spleen Pattern)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-CKKL-III
Record Dates: First submitted 2024-11-12; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Diarrhea-predominant Irritable Boewl Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Changkang granules (Experimental): 7.5g/bag, 1 bag per dose, 2 doses per day, oral，4 consecutive weeks.
  Interventions: Drug: Changkang granules
- Changkang granules Placebo (Placebo Comparator): 7.5g/bag, 1 bag per dose, 2 doses per day, oral，4 consecutive weeks.
  Interventions: Drug: Changkang Granules placebo

INTERVENTIONS:
Drug: Changkang granules — 7.5g/bag, 1 bag per dose, 2 doses per day, oral，4 consecutive weeks.
  Arms: Changkang granules
Drug: Changkang Granules placebo — 7.5g/bag, 1 bag per dose, 2 doses per day, oral，4 consecutive weeks.
  Arms: Changkang granules Placebo

SUMMARY:
This study will evaluate the efficacy and safety of Changkang granules in the treatment of irritable bowel syndrome with predominant Diarrhea ( Liver qi affecting the spleen pattern)

DETAILED DESCRIPTION:
This Randomized, Double-blind, Placebo-controlled, Multicenter Phase III clinical trial will evaluate the efficacy and safety of Changkang granules in the treatment of irritable bowel syndrome with predominant Diarrhea ( Liver qi affecting the spleen pattern)

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following inclusion criteria to be eligible for this trial:

  1. Age 18-65 years (inclusive), regardless of gender;
  2. Meet the Western medical diagnostic criteria for Irritable Bowel Syndrome with Predominant Diarrhea (Rome IV);
  3. Meet the Traditional Chinese Medicine diagnostic criteria for Liver qi affecting the spleen pattern
  4. Have a weekly average NRS score for abdominal pain ≥3.0 during the Run-In Period period, and have at least 2 days per week with stool form of type 6 or 7 (Bristol Stool Scale) during the Run-in period;
  5. Have an IBS-SSS score >175 at baseline;
  6. Have completed a colonoscopy within the past 12 months prior to the Run-in period, and meet one of the following conditions: ① Normal colonoscopy results with no organic changes; ② Abnormal colonoscopy report, such as hemorrhoids, polyps (diameter ≤5mm and number ≤3), etc., which the investigator determines can be included; ③ Previous colonoscopy report indicating polyps >5mm in diameter or >3 in number, which after endoscopic treatment 6 months ago, residual polyps are ≤5mm in diameter and ≤3 in number, and the investigator determines can be included;
  7. Voluntarily sign the informed consent form, and from the time of signing the informed consent form until the end of the last visit of the trial, the participant voluntarily accepts health education and maintains their usual diet and lifestyle, such as not changing dietary structure or exercise patterns.

Exclusion Criteria:

* Subjects with any of the following conditions are not eligible for enrollment in this study:

  1. Subjects who have less than 3 spontaneous bowel movements per week during the run-in period; or at least 2 days per week during the run-in period with stool consistency classified as type 1 or 2 on the Bristol Stool Scale;
  2. Patients with a history of severe mental or psychological disorders, or those scoring ≥63 on the Self-Rating Depression Scale (SDS), or ≥60 on the Self-Rating Anxiety Scale (SAS) during the screening period;
  3. Patients with a confirmed history of organic gastrointestinal diseases, including both gastrointestinal and non-gastrointestinal digestive system diseases, such as chronic superficial gastritis with erosions or bleeding of grade II or higher, chronic atrophic gastritis, peptic ulcers, inflammatory bowel disease, intestinal tuberculosis, intestinal ulcers, intestinal obstruction, intestinal adhesions, eosinophilic gastroenteritis, cholelithiasis with recurrent cholecystitis (patients with gallstones or gallbladder polyps ≤0.5 cm in diameter and no significant symptoms may be exempted from exclusion upon investigator's judgment), tuberculous peritonitis, liver cirrhosis, and digestive system tumors, etc.;
  4. Patients diagnosed with other diseases that affect the evaluation of abdominal pain and diarrhea, such as diarrhea caused by lactose intolerance, diarrhea after cholecystectomy, abdominal pain due to endometriosis, abdominal pain caused by hepatic and biliary stones or cholecystitis, abdominal pain due to chronic pancreatitis, etc.;
  5. Patients with a history of systemic diseases affecting gastrointestinal function, such as diabetes mellitus, hyperthyroidism or hypothyroidism, chronic renal insufficiency, autoimmune diseases (such as allergic colitis, allergic purpura, Behcet's syndrome, systemic lupus erythematosus), etc.;
  6. Patients with a history of major abdominal surgery involving the gastrointestinal tract, liver, gallbladder, spleen, or pancreas (subjects who have undergone appendectomy or cesarean section without impact on gut function may be exempted from exclusion upon investigator's judgment);
  7. Patients with unexplained recurrent positive fecal occult blood, unintentional weight loss, anemia, fever, or jaundice prior to screening;
  8. Abnormal liver function at baseline (ALT or AST >1.5 times the upper limit of normal) or abnormal renal function at baseline (Cr >upper limit of normal);
  9. Patients with a history of severe diseases in the respiratory, cardiovascular, cerebral, hepatic, renal, endocrine, immune, hematopoietic systems, as well as tumors and neurological diseases, deemed unsuitable for participation in this trial by the investigator;
  10. Patients who have used prokinetic agents, anticholinergic drugs, calcium channel blockers (excluding antihypertensive drugs), 5-HT3 receptor antagonists, antidiarrheals, antidepressants, anxiolytics, probiotics, analgesics, laxatives, etc., within 4 weeks before randomization;
  11. Patients who took rescue medication (piroxicam) during the run-in period;
  12. Pregnant or breastfeeding women, or those planning to conceive within 1 month after enrollment until the end of the trial;
  13. Patients suspected or known to be allergic to the investigational drug, rescue medication, or its components;
  14. Patients suspected or known to have a history of alcohol or drug abuse;
  15. Patients who participated in another interventional clinical trial and took investigational drugs within 1 month before screening;
  16. Patients whom the investigator deems unsuitable for clinical trial participation for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2026-11-11 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
abdominal pain response rate | 4 week
  The primary efficacy endpoint is the weekly response rate to abdominal pain after 4 weeks of treatment.

SECONDARY OUTCOMES:
The change in the average weekly score of abdominal pain compared to baseline | Baseline, Week 1，Week 2，week3 and week4
  Starting from the import period, subject diary cards will be collected, and the subjects will rate the "most severe abdominal pain in the past 24 hours" daily. The non empty diary card information of the subjects in the random first 7 days of the import period will be used as the baseline. Calculate the average weekly abdominal pain compared to baseline.
Weekly Composite Response Rate | 4 week
  Calculate the proportion of subjects with composite responses over a 4-week period. The intensity of abdominal pain and stool characteristics were obtained from diary cards, with non empty diary card information from participants in the first 7 days of randomization as the baseline. Effective subjects are defined as those who simultaneously meet the following efficacy criteria for at least 50% of the observation period.
The change in total IBS-SSS score and each individual item score from baseline | 4 week
  Irritable bowel syndrome symptom severity scale(IBS-SSS)is a scale to assess the severity of illness in patients with irritable bowel syndrome.The scale has a total score of 500, with a minimum score of 0. Higher scores indicate more severe IBS-related symptoms.The IBS-SSS scale includes an evaluation of five dimensions: degree of abdominal pain, frequency of abdominal pain and bloating, satisfaction with bowel movements, and impact on quality of life (Appendix 2). The total IBS-SSS scores and changes in each dimension from baseline were compared between the two groups.
The change in total IBS-SSS score and each individual item score from baseline | up to 10 week
  Irritable bowel syndrome symptom severity scale(IBS-SSS)is a scale to assess the severity of illness in patients with irritable bowel syndrome.The scale has a total score of 500, with a minimum score of 0. Higher scores indicate more severe IBS-related symptoms.The IBS-SSS scale includes an evaluation of five dimensions: degree of abdominal pain, frequency of abdominal pain and bloating, satisfaction with bowel movements, and impact on quality of life (Appendix 2).Calculate the total IBS-SSS scores at 3 and 6 weeks after discontinuation, as well as the changes in scores for each dimension compared to baseline.
Weekly stool consistency response rate | 4 week
  Fecal trait responders are defined as subjects who meet the efficacy criteria for fecal trait during at least 50% of the observation period (with at least one reduction of at least 50% in the number of days with type 6 or 7 fecal trait compared to baseline per week), and whose abdominal pain intensity remains unchanged or has improved.
The change in the number of days with stool type 6/7 compared to the baseline | Baseline,Week1,Week2,Week3 and Week4
  Compare the changes in the number of days with 6/7 bowel movements per week during the treatment period compared to baseline.
The change in the number of stool type 6/7 compared to baseline | Baseline, Week 1，Week 2，week3 and week4
  Compare the changes in the frequency of bowel movements of type 6/7 per week during the treatment period compared to baseline.
The changes in traditional chinese medicine syndrome score from baseline | 4 week
  Researchers used the IBS-D Liver Qi Multiplying Spleen Syndrome Scale to ask participants about traditional Chinese medicine syndrome related questions, fill out the scale, calculate the total score, and compare the changes in traditional Chinese medicine syndrome scores from baseline over the course of 4 weeks; Simultaneously calculate the change in TCM syndrome score from baseline for 2 weeks.The minimum score is 0 points, and the maximum score is 27 points. The higher the score, the worse it is.
The proportion of subjects with effective improvement in TCM syndrome score | 4 week
  Calculate the proportion of subjects who have effectively improved their TCM syndrome score over a period of 4 weeks.
The change in the score of individual item of TCM symptoms compared to baseline | 4 week
  Compare the changes in individual symptom scores of traditional Chinese medicine over a 4-week period compared to baseline.
The decrease percentage of individual TCM symptoms compared to baseline | 4 week
  Compare the percentage decrease of individual symptoms in traditional Chinese medicine over a period of 4 weeks.

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Baoding First Traditional Chinese Medicine Hospital, Baoding
  - No. 5, Beixiange Street, Xuanwu District, Beijing, Beijing
  - The Second Affiliated Hospital of Hunan University of Chinese Medicine, Changsha
  - Changde Second People's Hospital, Chengde
  - Chengdu Shuangliu District First People's Hospital, Chengdu
  - Sichuan University West China Hospital, Chengdu
  - Guangzhou First People's Hospital, Guangzhou
  - Zhejiang Provincial Tongde Hospital, Hangzhou
  - Zhejiang Xinhua Hospital, Hangzhou
  - Kaifeng City Traditional Chinese Medicine Hospital, Kaifeng
  - Gansu Provincial Hospital of Traditional Chinese Medicine, Lanzhou
  - Luoyang Central Hospital, Luoyang
  - Luoyang First People's Hospital, Luoyang
  - Jiangxi University of Traditional Chinese Medicine Affiliated Hospital, Nanchang
  - Nanjing Traditional Chinese Medicine Hospital, Nanjing
  - Guangxi Traditional Chinese Medicine University Affiliated Rui Kang Hospital, Nanning
  - Sanmenxia Central Hospital, Sanmenxia
  - Shanghai University of Traditional Chinese Medicine Affiliated Longhua Hospital, Shanghai
  - Liaoning University of Traditional Chinese Medicine Third Affiliated Hospital, Shenyang
  - Hebei Provincial Hospital of Traditional Chinese Medicine, Shijiazhuang
  - Hebei Provincial People's Hospital, Shijiazhuang
  - Tianjin University of Traditional Chinese Medicine Second Affiliated Hospital, Tianjin
  - Wenzhou Medical University Affiliated Second Hospital, Wenzhou
  - Wenzhou Traditional Chinese Medicine Hospital, Wenzhou
  - Huazhong University of Science and Technology Tongji Medical College Affiliated Union Hospital, Wuhan
  - Hubei Provincial Hospital of Traditional Chinese Medicine, Wuhan
  - Shanxi Provincial Hospital of Traditional Chinese Medicine, Xi'an
  - Shanxi University of Chinese Medicine Affiliated Hospital, Xianyang
  - The Second Affiliated Hospital of Shanxi University of Chinese Medicine, Xianyang
  - Yangquan Coal Industry (Group) Co., Ltd. General Hospital, Yangquan